CLINICAL TRIAL: NCT02016209
Title: Phase II Study of Neoadjuvant Chemotherapy of Nanoparticle Albumin-bound Paclitaxel Plus Carboplatin/Cisplatin in Stage Ⅱ B and IIIA Non-small Cell Lung Cancer Patients
Brief Title: Neoadjuvant Chemotherapy of Nanoparticle Albumin-bound Paclitaxel in Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Qiong Zhao, Chief of Department of Thoracic Oncology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYTOP1402
Record Dates: First submitted 2013-12-07; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Taxes; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nanoparticle albumin-bound paclitaxel (Experimental): Neoadjuvant chemotherapy of platinum-based nanoparticle albumin-bound paclitaxel in stage Ⅱ B and IIIA non-small cell lung cancer
  Interventions: Drug: nanoparticle albumin-bound paclitaxel

INTERVENTIONS:
Drug: nanoparticle albumin-bound paclitaxel — Neoadjuvant chemotherapy of nanoparticle albumin-bound paclitaxel in stage Ⅱ B and IIIA non-small cell lung cancer
  Other Names: nab-paclitaxel

SUMMARY:
platinum-based albumin-bound paclitaxel regimen in advanced non-small cell lung cancer (NSCLC) especially in lung squamous cell carcinoma has a better tumor response rate and safety than solvent-based paclitaxel.However, the safety and efficacy is uncertain in neoadjuvant therapy.

DETAILED DESCRIPTION:
The main purpose of this study is to observe the safety and efficacy of platinum-based albumin-bound paclitaxel regimen in the treatment of non-small cell lung cancer (NSCLC) of stage Ⅱ B and IIIA .

ELIGIBILITY:
Inclusion Criteria:

1.Histological or cytological diagnosis of NSCLC of Stage Ⅱ B and IIIA .

2.18 years or older 3.Performance Status 0 to 2; 4.Appraisable disease; 5.patients can tolerant chemotherapy; 6.Total bilirubin 1.5 x upper limit of normal (ULN); 7.Creatinine clearance 60ml/min (calculated according to Cockcroft-gault formula).

Exclusion Criteria:

1.Any systemic anticancer treatment for NSCLC；2.Local radiotherapy for NSCLC；3.In this study within five years prior to the start of treatment with other than NSCLC patients with other cancers.4.Any instability in systemic disease; 5.Allergic to paclitaxel or Platinum;6.Pregnant or lactating women;7.Other researchers believe that does not fit into the group

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate and Number of Adverse Events | From date of randomization until the date of progression, assessed up to 2 months

SECONDARY OUTCOMES:
disease free survival | From date of surgery until the date of first documented progression, assessed up to 36 months

OTHER OUTCOMES:
dynamic circulating tumor cell changes during treatment | baseline, 3 weeks and up to progression disease

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Zhao, PhD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The first affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China